CLINICAL TRIAL: NCT00280293
Title: A Randomized, Double-blind, Placebo-controlled, Trial of Lamotrigine add-on Therapy in Outpatients With Bipolar Disorder, Depressed or Mixed Phase and Cocaine Dependence
Brief Title: Lamotrigine add-on Therapy for Bipolar Disorder and Cocaine Dependency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, Principal Investigator, MD/PhD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05T-704
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-07

CONDITIONS: Bipolar Disorder; Cocaine Dependence
Keywords: Bipolar Disorder; Cocaine Dependence; Dual Diagnosis
MeSH Terms: conditions — Bipolar Disorder; Cocaine-Related Disorders | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): LAmotrigine
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine
  Arms: 2
Drug: Placebo — Placebo
  Arms: 1

SUMMARY:
The purpose of this study is to determine if lamotrigine add-on therapy is associated with decreased cocaine craving and improvement in depressive symptom severity than placebo in a group of outpatients with bipolar disorder and cocaine dependence. Additionally, this study is examining whether lamotrigine add-on therapy is associated with decreased cocaine use and the improvement of manic symptom severity than placebo in a group of outpatients with bipolar disorder and cocaine dependence.

DETAILED DESCRIPTION:
One hundred and twenty (120) adult outpatients with bipolar I, II, not otherwise specified, or cyclothymic disorder and current cocaine dependence will be enrolled. After obtaining informed consent baseline assessment measures will be administered including the Structured Clinical Interview for Diagnostic Statistical Manual-IV Axis I Disorders. Drug use will be assessed using the timeline-followback method to quantify days and amount of drug use, urine drug screens will also be obtained and craving will be assessed with the Cocaine Craving Questionnaire. Mood symptoms will be quantified at each weekly visit with the Hamilton Rating Scale for Depression (17-item version), Quick Inventory of Depressive Symptomatology-SR (QIDS-SR), and Young Mania Rating Scale (YMRS). Impulsivity will be assessed at weeks 0, 5 and 10 with the Barratt Impulsiveness Scale (BIS, Barratt et al 1983). Cognition will be assessed at weeks 0, 5, and 10 with the Rey Auditory Verbal Learning Test (RAVLT) and STROOP color-word task. The Addiction Severity Index (ASI) will be administered at baseline and week 10. The Psychobiology of Recovery in Depression-III Somatic Symptom Scale (PRD-III)will be administered every 2 weeks to track side effects. A study psychiatrist will assess participant-reported side effects weekly. Women of childbearing age will be given a test to rule out pregnancy. Subjects will be randomized and Lamotrigine therapy or identical appearing placebo add-on therapy in a double- blind fashion will be initiated at 25 mg/day and increased to 200 mg/day using a slow upward titration over 5 weeks (as outlined by Calabrese et al 2000 and following the package insert) to minimize risk of side effects such as rash. After that time additional increases in 100 mg/day increments to a maximum of 400 mg/day can be made if the medication is well tolerated and HRSD scores have decreased by ≤ 40% from baseline or Cocaine Craving Questionaire (CCQ) scores have decreased ≤ 25% from baseline or participants continue to use cocaine in past week based on either self-report or urine drug screen results. Subjects will be assessed weekly for mood and drug use/craving and every four weeks for cognition over 10 weeks. All of the assessments may be provided in Spanish, if needed. Additionally, a Spanish-speaking research assistant and study psychiatrist will be available at all times.

Subjects will be paid $30 for each visit and given $2 restaurant coupons. Parking tokens ($3) or bus passes ($2) will also be provided. Concomitant medications will be managed with an algorithm that discourages but, if necessary, allows changes in other psychiatric medications. At the completion of 10 weeks of blinded therapy participants in both groups will be offered 4 weeks of open-label therapy either continuing at the week 10 dose in those on active medication or slowly titrated upward for those on placebo. Participants will be assessed with the HRSD, QIDS-SR, YMRS, CCQ and drug use quantified at biweekly appointments with the RAVLT and STROOP also administered at week 14 exit. Participants will not be paid for participation in the open-label phase but bus tokens and parking passes will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar I, II, not otherwise specified or cyclothymic disorders
* Currently depressed or mixed mood state
* Ages 18-70 years
* Men or women
* Self-reported cocaine use within 14 days prior to randomization
* English or Spanish speaking
* Baseline Hamilton Depression Rating Scale (HRSD17) score ≥ 10

Exclusion Criteria:

* Currently taking an enzyme inducing or inhibiting anticonvulsant (e.g. valproic acid, carbamazepine)
* Current severe psychotic features (e.g. daily auditory hallucinations, fixed delusions, severely disorganized thought processes) that require antipsychotic therapy, and that do not appear to be secondary to cocaine use
* Active suicidal ideation (plan and intent) or ≥2 attempts in past 12 months or any attempt in the past month
* Highly unstable medical condition
* Change in concomitant psychiatric medications (e.g. initiated antipsychotic) or in other substance abuse treatment (e.g. began intensive outpatient treatment) within 7 days prior to study entry
* Vulnerable populations (e.g. pregnant or nursing women, prisoners, mentally retarded)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, M.D., Ph.D., Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 112 participants with at least one post-baseline visit were recruited between 2006 and 2010 at our research clinic in Dallas, TX and included for analysis.
Pre-assignment Details: Participants with a diagnosis of bipolar I, II or NOS disorders currently depressed or mixed mood with current cocaine dependence and self-reported use within 14 days were included. The study drug was added to existing psychiatric medications or given as monotherapy when participants were not taking other medications at baseline.
Groups:
- Lamotrigine: Lamotrigine therapy was initiated at 25 mg/day and increased to 200 mg/day using a slow upward titration over 5 weeks. After that time additional increases in 100 mg/day increments to a maximum of 400 mg/day were made if the medication was well tolerated and signs of poor response were noted.
- Placebo: Placebo group received medication in identical color/sizes as the lamotrigine group. Placebo therapy was initiated at 25 mg/day and increased to 200 mg/day using a slow upward titration over 5 weeks. After that time additional increases in 100 mg/day increments to a maximum of 400 mg/day were made if the medication was well tolerated and signs of poor response were noted.
Period: Overall Study
Arm/Group | Lamotrigine | Placebo
Started | 55 | 57
Completed | 29 | 34
Not Completed | 26 | 23
Not completed — Protocol Violation | 3 | 0
Not completed — Physician Decision | 5 | 4
Not completed — Lost to Follow-up | 14 | 12
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Incarceration/Legal Reasons | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine | Placebo | Total
Number analyzed (Participants) | 55 | 57 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 57 | 112
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.1 (7.3) | 43.5 (10.0) | 44.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 32 | 35 | 67
Region of Enrollment [Number; unit: participants]
  United States | 55 | 57 | 112

OUTCOME MEASURES:

1. Primary Outcome: Days of Cocaine Use
Description: Number of days of cocaine use during the 7 days that comprise week 10 of the protocol, by self report, or at last assessment if participant withdrew early, as assessed by the Timeline Followback method.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 55 | 57
days | 1.8 (2.0) | 2.8 (4.0)

2. Secondary Outcome: Depression Score on the Hamilton Rating Scale For Depression
Description: Total score on the Hamilton Rating Scale for Depression at week 10 visit or at last assessment if participant withdrew early(total score values range 0 - 52. A higher score indicates more severe depression.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 55 | 57
units on a scale | 13.4 (8.5) | 13.6 (8.2)

3. Secondary Outcome: Dollars Spent
Description: Dollars spent on cocaine during the 7 days of week 10, or at last assessment if participant withdrew early, based on self report.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 55 | 57
Dollars | 68.6 (121.1) | 155.4 (355.5)

4. Primary Outcome: Positive Urine Drug Screens
Description: Percentage of participants with a positive urine drug screen for cocaine at the week 10 visit or at last assessment if participant withdrew early.
Time Frame: 10 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 55 | 57
percentage of participants | 67.3 | 73.6

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study between 2006 and 2010. Each participant was enrolled for 10 weeks. Adverse events were collected for the full 10 weeks, beginning after consent was signed.
Description: Adverse events were assessed by a weekly questionnaire at each appointment.
Arm/Group | Lamotrigine | Placebo
Serious Adverse Events (participants affected / at risk) | 5/55 | 4/57
Other Adverse Events (participants affected / at risk) | 6/55 | 4/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lamotrigine (N=55) | Placebo (N=57)
Inpatient psychiatric admittance (Psychiatric disorders) | 3 (3) | 1 (1) — For suicidal ideation/plan/intent
Inpatient admittance for blood transfusion (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — Due to congenital Sickle Cell Anemia
Inpatient admittance for urinary tract blockage (Renal and urinary disorders) | 0 (0) | 1 (1) — Due to pre-existing benign tumors
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Inpatient admittance due to hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Fall related injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Expression of violent thoughts/ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lamotrigine (N=55) | Placebo (N=57)
Admittance to psychiatric facility (Psychiatric disorders) | 1 (1) | 0 (0) — As terms for violating parole (for a positive cocaine UDS)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma attack (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Nosebleed (Vascular disorders) | 1 (1) | 0 (0)
Superficial Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cut related injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall related injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abscessed Tooth (Infections and infestations) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The weekly UDS (rather than thrice weekly as is customary in cocaine trials) design feature decreased our number of observations and statistical power, and did not provide us with a complete picture of cocaine use between weekly visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less